CLINICAL TRIAL: NCT03683394
Title: Multidomain Alzheimers Risk Reduction Study (MARRS) Pilot
Brief Title: Systematic Multi-domain Alzheimer's Risk Reduction Trial
Acronym: SMARRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01AG057508 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-25 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Dementia; Alzheimer Disease
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Participants will be randomized after baseline assessments to the SMARRT intervention arm or Health Education (HE) control arm. Randomization will be stratified by clinic, race/ethnicity (non-Hispanic white vs. non-white or Hispanic) and age (70-79, 80-89).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMARRT Intervention (Active Comparator): The SMARRT intervention team will use a standardized procedure to develop an individualized Alzheimer's risk profile for each participant randomized to the SMARRT intervention arm. Participants will then meet in-person with an interventionist to review their risk profile and develop an initial personalized risk reduction action plan. For the few participants enrolled during COVID, initial interventionist visits were conducted by phone. Targeted areas will include: increasing physical, mental and social activities; quitting smoking; healthy diet; controlling cardiovascular risk factors (diabetes, hypertension), including avoiding hypoglycemia in people with diabetes; reducing depressive symptoms; improving sleep; and decreasing use of potentially harmful medications.
  Interventions: Behavioral: SMARRT Intervention
- Health Education Intervention (Active Comparator): Participants in the Health Education arm will be mailed general information that will address factors that will be targeted in the SMARRT intervention, including physical, mental and social engagement; management of cardiovascular risk factors; quitting smoking, healthy diet; depression; sleep; and contraindicated medications. HE participants will not be provided with personalized information about their risk of Alzheimer's and dementia.
  Interventions: Behavioral: Health Education Intervention

INTERVENTIONS:
Behavioral: SMARRT Intervention — Interventionists will follow a standard protocol for delivering the SMARRT intervention that allows for personalization of the specific risk reduction action plan; these plans will evolve over time according to participant progress, motivation and preferences or newly identified risk factors. Staff will use a tracking database to record information for each participant, including session dates, identified risk factors, motivational barriers and important values, and the outcome of discussions around developing goals. For each participant, the exact number and mode (phone or in-person) of contacts will differ, but we will aim to have at least 1 contact per month with each participant. Best practice will include in-person meetings twice a year during the 2-year intervention period.
  Arms: SMARRT Intervention
Behavioral: Health Education Intervention — Participants randomized to the Health Education (HE) group will receive mailed materials (typically 1-2 pages) every 3 months. This will include general information on Alzheimer's and dementia risk reduction using materials from sources such as the Alzheimer's Association and educational materials commonly provided as part of routine care at Kaiser Permanente Washington (KPWA).
  Arms: Health Education Intervention

SUMMARY:
The primary goal of this randomized controlled trial (RCT) is to pilot-test a personalized, pragmatic, multi-domain Alzheimer's disease risk reduction intervention in a U.S. integrated healthcare delivery system.

DETAILED DESCRIPTION:
We propose to randomize 200 higher-risk older adults (age 70-89 with low-normal performance on cognitive testing and 2+ modifiable risk factors that will be targeted by our intervention) to a two-year Systematic Multi-Domain Alzheimer's Risk Reduction Trial (SMARRT) intervention or a Health Education (HE) control.

The SMARRT team will work with participants randomized to the intervention arm to develop a tailored action plan to address risk reduction. Targeted areas will include: increasing physical, mental and social activities; controlling cardiovascular risk factors (diabetes, hypertension); quitting smoking; reducing depressive symptoms; improving sleep; neuroprotective diet; and decreasing use of potentially harmful medications. HE participants will receive periodic handouts on these topics by mail.

Changes made to the protocol due to COVID-19, i.e. switching to telephone data collection, will likely limit our ability to examine cognitive change effectively, as several of the most important cognitive tests cannot be administered via telephone.

ELIGIBILITY:
Inclusion Criteria:

* 70-89 Years of Age
* Fluent in the English Language
* Low-normal performance on a brief telephone cognitive screen, measured using the Cognitive Abilities Screening Instruments (CASI). Low-normal scores are defined as 26-29.
* Has at least two additional risk factors that will be targeted by the intervention.

Exclusion Criteria:

* Residing in a skilled nursing or rehabilitation facility
* Receiving palliative care or hospice services
* Charlson comorbidity index score of greater than 5
* Bipolar illness or schizophrenia
* Current alcohol or drug use disorder
* Receiving chronic opioid therapy
* Parkinson's disease, amyotrophic lateral sclerosis, or multiple sclerosis
* Severe visual or hearing impairment
* Requests not to be contacted or not to have their medical record reviewed for research
* Prior evidence of dementia

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 172 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Dublin, MD, PhD, Principal Investigator — Kaiser Permanente; Kristine Yaffe, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Kaiser Permanente Washington Health Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer's Disease International. World Alzheimer Report 2015: The Global Impact of Dementia, An Analysis of Prevalence, Incidence, Cost and Trends. London: Alzheimer's Disease International (ADI); 2015.
- [Background] Alzheimer's Association. 2011 Alzheimer's disease facts and figures. Alzheimers Dement. 2011 Mar;7(2):208-44. doi: 10.1016/j.jalz.2011.02.004. PMID 21414557
- [Background] Atri A, Frolich L, Ballard C, Tariot PN, Molinuevo JL, Boneva N, Windfeld K, Raket LL, Cummings JL. Effect of Idalopirdine as Adjunct to Cholinesterase Inhibitors on Change in Cognition in Patients With Alzheimer Disease: Three Randomized Clinical Trials. JAMA. 2018 Jan 9;319(2):130-142. doi: 10.1001/jama.2017.20373. PMID 29318278
- [Background] Bezprozvanny I. The rise and fall of Dimebon. Drug News Perspect. 2010 Oct;23(8):518-23. doi: 10.1358/dnp.2010.23.8.1500435. PMID 21031168
- [Background] Cummings JL, Morstorf T, Zhong K. Alzheimer's disease drug-development pipeline: few candidates, frequent failures. Alzheimers Res Ther. 2014 Jul 3;6(4):37. doi: 10.1186/alzrt269. eCollection 2014. PMID 25024750
- [Background] Fagan T. Clinical Trials of Intravenous Bapineuzumab Halted. Alzheimer Research Forum onlineAugust 8, 2012.
- [Background] Fagan T. Lilly Halts IDENTITY Trials as Patients Worsen on Secretase Inhibitor. Alzheimer Research Forum onlineAugust 18, 2010.
- [Background] Honig LS, Vellas B, Woodward M, Boada M, Bullock R, Borrie M, Hager K, Andreasen N, Scarpini E, Liu-Seifert H, Case M, Dean RA, Hake A, Sundell K, Poole Hoffmann V, Carlson C, Khanna R, Mintun M, DeMattos R, Selzler KJ, Siemers E. Trial of Solanezumab for Mild Dementia Due to Alzheimer's Disease. N Engl J Med. 2018 Jan 25;378(4):321-330. doi: 10.1056/NEJMoa1705971. PMID 29365294
- [Background] Jeffrey S. IVIG Fails in Phase 3 for Alzheimer's. Medscape Today May 7, 2013.
- [Background] Salloway S, Sperling R, Fox NC, Blennow K, Klunk W, Raskind M, Sabbagh M, Honig LS, Porsteinsson AP, Ferris S, Reichert M, Ketter N, Nejadnik B, Guenzler V, Miloslavsky M, Wang D, Lu Y, Lull J, Tudor IC, Liu E, Grundman M, Yuen E, Black R, Brashear HR; Bapineuzumab 301 and 302 Clinical Trial Investigators. Two phase 3 trials of bapineuzumab in mild-to-moderate Alzheimer's disease. N Engl J Med. 2014 Jan 23;370(4):322-33. doi: 10.1056/NEJMoa1304839. PMID 24450891
- [Background] Larson EB, Yaffe K, Langa KM. New insights into the dementia epidemic. N Engl J Med. 2013 Dec 12;369(24):2275-7. doi: 10.1056/NEJMp1311405. Epub 2013 Nov 27. No abstract available. PMID 24283198
- [Background] Yaffe K. Modifiable Risk Factors and Prevention of Dementia: What Is the Latest Evidence? JAMA Intern Med. 2018 Feb 1;178(2):281-282. doi: 10.1001/jamainternmed.2017.7299. No abstract available. PMID 29255907
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Norton S, Matthews FE, Barnes DE, Yaffe K, Brayne C. Potential for primary prevention of Alzheimer's disease: an analysis of population-based data. Lancet Neurol. 2014 Aug;13(8):788-94. doi: 10.1016/S1474-4422(14)70136-X. PMID 25030513
- [Background] Langa KM, Larson EB, Crimmins EM, Faul JD, Levine DA, Kabeto MU, Weir DR. A Comparison of the Prevalence of Dementia in the United States in 2000 and 2012. JAMA Intern Med. 2017 Jan 1;177(1):51-58. doi: 10.1001/jamainternmed.2016.6807. PMID 27893041
- [Background] Manton KC, Gu XL, Ukraintseva SV. Declining prevalence of dementia in the U.S. elderly population. Adv Gerontol. 2005;16:30-7. PMID 16075674
- [Background] Matthews FE, Arthur A, Barnes LE, Bond J, Jagger C, Robinson L, Brayne C; Medical Research Council Cognitive Function and Ageing Collaboration. A two-decade comparison of prevalence of dementia in individuals aged 65 years and older from three geographical areas of England: results of the Cognitive Function and Ageing Study I and II. Lancet. 2013 Oct 26;382(9902):1405-12. doi: 10.1016/S0140-6736(13)61570-6. Epub 2013 Jul 17. PMID 23871492
- [Background] Qiu C, von Strauss E, Backman L, Winblad B, Fratiglioni L. Twenty-year changes in dementia occurrence suggest decreasing incidence in central Stockholm, Sweden. Neurology. 2013 May 14;80(20):1888-94. doi: 10.1212/WNL.0b013e318292a2f9. Epub 2013 Apr 17. PMID 23596063
- [Background] Rocca WA, Petersen RC, Knopman DS, Hebert LE, Evans DA, Hall KS, Gao S, Unverzagt FW, Langa KM, Larson EB, White LR. Trends in the incidence and prevalence of Alzheimer's disease, dementia, and cognitive impairment in the United States. Alzheimers Dement. 2011 Jan;7(1):80-93. doi: 10.1016/j.jalz.2010.11.002. PMID 21255746
- [Background] Schrijvers EM, Verhaaren BF, Koudstaal PJ, Hofman A, Ikram MA, Breteler MM. Is dementia incidence declining?: Trends in dementia incidence since 1990 in the Rotterdam Study. Neurology. 2012 May 8;78(19):1456-63. doi: 10.1212/WNL.0b013e3182553be6. Epub 2012 May 2. PMID 22551732
- [Background] Wu YT, Beiser AS, Breteler MMB, Fratiglioni L, Helmer C, Hendrie HC, Honda H, Ikram MA, Langa KM, Lobo A, Matthews FE, Ohara T, Peres K, Qiu C, Seshadri S, Sjolund BM, Skoog I, Brayne C. The changing prevalence and incidence of dementia over time - current evidence. Nat Rev Neurol. 2017 Jun;13(6):327-339. doi: 10.1038/nrneurol.2017.63. Epub 2017 May 12. PMID 28497805
- [Background] Lee KS, Lee Y, Back JH, Son SJ, Choi SH, Chung YK, Lim KY, Noh JS, Koh SH, Oh BH, Hong CH. Effects of a multidomain lifestyle modification on cognitive function in older adults: an eighteen-month community-based cluster randomized controlled trial. Psychother Psychosom. 2014;83(5):270-8. doi: 10.1159/000360820. Epub 2014 Aug 6. PMID 25116574
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Rosenberg A, Ngandu T, Rusanen M, Antikainen R, Backman L, Havulinna S, Hanninen T, Laatikainen T, Lehtisalo J, Levalahti E, Lindstrom J, Paajanen T, Peltonen M, Soininen H, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Solomon A, Kivipelto M. Multidomain lifestyle intervention benefits a large elderly population at risk for cognitive decline and dementia regardless of baseline characteristics: The FINGER trial. Alzheimers Dement. 2018 Mar;14(3):263-270. doi: 10.1016/j.jalz.2017.09.006. Epub 2017 Oct 19. PMID 29055814
- [Background] Andrieu S, Guyonnet S, Coley N, Cantet C, Bonnefoy M, Bordes S, Bories L, Cufi MN, Dantoine T, Dartigues JF, Desclaux F, Gabelle A, Gasnier Y, Pesce A, Sudres K, Touchon J, Robert P, Rouaud O, Legrand P, Payoux P, Caubere JP, Weiner M, Carrie I, Ousset PJ, Vellas B; MAPT Study Group. Effect of long-term omega 3 polyunsaturated fatty acid supplementation with or without multidomain intervention on cognitive function in elderly adults with memory complaints (MAPT): a randomised, placebo-controlled trial. Lancet Neurol. 2017 May;16(5):377-389. doi: 10.1016/S1474-4422(17)30040-6. Epub 2017 Mar 27. PMID 28359749
- [Background] Lam LC, Chan WC, Leung T, Fung AW, Leung EM. Would older adults with mild cognitive impairment adhere to and benefit from a structured lifestyle activity intervention to enhance cognition?: a cluster randomized controlled trial. PLoS One. 2015 Mar 31;10(3):e0118173. doi: 10.1371/journal.pone.0118173. eCollection 2015. PMID 25826620
- [Background] Moll van Charante EP, Richard E, Eurelings LS, van Dalen JW, Ligthart SA, van Bussel EF, Hoevenaar-Blom MP, Vermeulen M, van Gool WA. Effectiveness of a 6-year multidomain vascular care intervention to prevent dementia (preDIVA): a cluster-randomised controlled trial. Lancet. 2016 Aug 20;388(10046):797-805. doi: 10.1016/S0140-6736(16)30950-3. Epub 2016 Jul 26. PMID 27474376
- [Background] Teng EL, Hasegawa K, Homma A, Imai Y, Larson E, Graves A, Sugimoto K, Yamaguchi T, Sasaki H, Chiu D, et al. The Cognitive Abilities Screening Instrument (CASI): a practical test for cross-cultural epidemiological studies of dementia. Int Psychogeriatr. 1994 Spring;6(1):45-58; discussion 62. doi: 10.1017/s1041610294001602. PMID 8054493
- [Background] Kukull WA, Higdon R, Bowen JD, McCormick WC, Teri L, Schellenberg GD, van Belle G, Jolley L, Larson EB. Dementia and Alzheimer disease incidence: a prospective cohort study. Arch Neurol. 2002 Nov;59(11):1737-46. doi: 10.1001/archneur.59.11.1737. PMID 12433261
- [Background] Corrada MM, Brookmeyer R, Paganini-Hill A, Berlau D, Kawas CH. Dementia incidence continues to increase with age in the oldest old: the 90+ study. Ann Neurol. 2010 Jan;67(1):114-21. doi: 10.1002/ana.21915. PMID 20186856
- [Background] Charlson M, Szatrowski TP, Peterson J, Gold J. Validation of a combined comorbidity index. J Clin Epidemiol. 1994 Nov;47(11):1245-51. doi: 10.1016/0895-4356(94)90129-5. PMID 7722560
- [Background] Kivipelto M, Solomon A, Ahtiluoto S, Ngandu T, Lehtisalo J, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Nissinen A, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H. The Finnish Geriatric Intervention Study to Prevent Cognitive Impairment and Disability (FINGER): study design and progress. Alzheimers Dement. 2013 Nov;9(6):657-65. doi: 10.1016/j.jalz.2012.09.012. Epub 2013 Jan 17. PMID 23332672
- [Background] Harrison J, Minassian SL, Jenkins L, Black RS, Koller M, Grundman M. A neuropsychological test battery for use in Alzheimer disease clinical trials. Arch Neurol. 2007 Sep;64(9):1323-9. doi: 10.1001/archneur.64.9.1323. PMID 17846273
- [Background] Harrison J, Rentz DM, McLaughlin T, Niecko T, Gregg KM, Black RS, Buchanan J, Liu E, Grundman M; ELN-AIP-901 Study Investigator Group. Cognition in MCI and Alzheimer's disease: baseline data from a longitudinal study of the NTB. Clin Neuropsychol. 2014;28(2):252-68. doi: 10.1080/13854046.2013.875595. Epub 2014 Feb 13. PMID 24521259
- [Background] Topolski TD, LoGerfo J, Patrick DL, Williams B, Walwick J, Patrick MB. The Rapid Assessment of Physical Activity (RAPA) among older adults. Prev Chronic Dis. 2006 Oct;3(4):A118. Epub 2006 Sep 15. PMID 16978493
- [Background] Hahn EA, Beaumont JL, Pilkonis PA, Garcia SF, Magasi S, DeWalt DA, Cella D. The PROMIS satisfaction with social participation measures demonstrated responsiveness in diverse clinical populations. J Clin Epidemiol. 2016 May;73:135-41. doi: 10.1016/j.jclinepi.2015.08.034. Epub 2016 Feb 27. PMID 26931288
- [Background] Vemuri P, Lesnick TG, Przybelski SA, Machulda M, Knopman DS, Mielke MM, Roberts RO, Geda YE, Rocca WA, Petersen RC, Jack CR Jr. Association of lifetime intellectual enrichment with cognitive decline in the older population. JAMA Neurol. 2014 Aug;71(8):1017-24. doi: 10.1001/jamaneurol.2014.963. PMID 25054282
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Barnes LL, Bennett DA, Aggarwal NT. MIND diet slows cognitive decline with aging. Alzheimers Dement. 2015 Sep;11(9):1015-22. doi: 10.1016/j.jalz.2015.04.011. Epub 2015 Jun 15. PMID 26086182
- [Background] Morris MC, Tangney CC, Wang Y, Sacks FM, Bennett DA, Aggarwal NT. MIND diet associated with reduced incidence of Alzheimer's disease. Alzheimers Dement. 2015 Sep;11(9):1007-14. doi: 10.1016/j.jalz.2014.11.009. Epub 2015 Feb 11. PMID 25681666
- [Background] Radloff LS. The CES-D scale: A self-report depression scale for research in the general population. Applied Psychological Measurement. 1977;1(3):385-401.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] By the American Geriatrics Society 2015 Beers Criteria Update Expert Panel. American Geriatrics Society 2015 Updated Beers Criteria for Potentially Inappropriate Medication Use in Older Adults. J Am Geriatr Soc. 2015 Nov;63(11):2227-46. doi: 10.1111/jgs.13702. Epub 2015 Oct 8. PMID 26446832
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Amariglio RE, Donohue MC, Marshall GA, Rentz DM, Salmon DP, Ferris SH, Karantzoulis S, Aisen PS, Sperling RA; Alzheimer's Disease Cooperative Study. Tracking early decline in cognitive function in older individuals at risk for Alzheimer disease dementia: the Alzheimer's Disease Cooperative Study Cognitive Function Instrument. JAMA Neurol. 2015 Apr;72(4):446-54. doi: 10.1001/jamaneurol.2014.3375. PMID 25706191
- [Background] Hays RD, Bjorner JB, Revicki DA, Spritzer KL, Cella D. Development of physical and mental health summary scores from the patient-reported outcomes measurement information system (PROMIS) global items. Qual Life Res. 2009 Sep;18(7):873-80. doi: 10.1007/s11136-009-9496-9. Epub 2009 Jun 19. PMID 19543809
- [Background] Petersen RC, Lopez O, Armstrong MJ, Getchius TSD, Ganguli M, Gloss D, Gronseth GS, Marson D, Pringsheim T, Day GS, Sager M, Stevens J, Rae-Grant A. Practice guideline update summary: Mild cognitive impairment [RETIRED]: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology. Neurology. 2018 Jan 16;90(3):126-135. doi: 10.1212/WNL.0000000000004826. Epub 2017 Dec 27. PMID 29282327
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Winblad B, Palmer K, Kivipelto M, Jelic V, Fratiglioni L, Wahlund LO, Nordberg A, Backman L, Albert M, Almkvist O, Arai H, Basun H, Blennow K, de Leon M, DeCarli C, Erkinjuntti T, Giacobini E, Graff C, Hardy J, Jack C, Jorm A, Ritchie K, van Duijn C, Visser P, Petersen RC. Mild cognitive impairment--beyond controversies, towards a consensus: report of the International Working Group on Mild Cognitive Impairment. J Intern Med. 2004 Sep;256(3):240-6. doi: 10.1111/j.1365-2796.2004.01380.x. PMID 15324367
- [Background] Cohen J. Statistical power analysis for the behavioral sciences (2nd ed). Hillsdale, N.J.: Lawrence Earlbaum Associates; 1988.
- [Background] Li C, Friedman B, Conwell Y, Fiscella K. Validity of the Patient Health Questionnaire 2 (PHQ-2) in identifying major depression in older people. J Am Geriatr Soc. 2007 Apr;55(4):596-602. doi: 10.1111/j.1532-5415.2007.01103.x. PMID 17397440
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Derived] Yaffe K, Vittinghoff E, Dublin S, Peltz CB, Fleckenstein LE, Rosenberg DE, Barnes DE, Balderson BH, Larson EB. Effect of Personalized Risk-Reduction Strategies on Cognition and Dementia Risk Profile Among Older Adults: The SMARRT Randomized Clinical Trial. JAMA Intern Med. 2024 Jan 1;184(1):54-62. doi: 10.1001/jamainternmed.2023.6279. PMID 38010725

RESULTS

PARTICIPANT FLOW:
Groups:
- SMARRT Intervention: The SMARRT intervention team used a standardized procedure to develop an individualized Alzheimer's risk profile for each participant randomized to the SMARRT intervention arm. Participants then met with an interventionist to review their risk profile and develop an initial personalized risk reduction action plan. Targeted areas included: increasing physical, mental and social activities; quitting smoking; healthy diet; controlling cardiovascular risk factors (diabetes, hypertension), including avoiding hypoglycemia in people with diabetes; reducing depressive symptoms; improving sleep; and decreasing use of potentially harmful medications.
  SMARRT Intervention: Interventionists will follow a standard protocol for delivering the SMARRT intervention that allows for personalization of the specific risk reduction action plan; these plans will evolve over time according to participant progress, motivation and preferences or newly identified risk factors. Staff will use a tracking database to record information for each participant, including session dates, identified risk factors, motivational barriers and important values, and the outcome of discussions around developing goals. For each participant, the exact number and mode (phone or in-person) of contacts will differ, but we will aim to have at least 1 contact per month with each participant. Best practice will include in-person meetings twice a year during the 2-year intervention period.
- Health Education Control: Participants in the Health Education arm were mailed general information that addressed factors targeted in the SMARRT intervention, including physical, mental and social engagement; management of cardiovascular risk factors; quitting smoking, healthy diet; depression; sleep; and contraindicated medications. HE participants were not provided with personalized information about their risk of Alzheimer's and dementia.
  Health Education Intervention: Participants randomized to the Health Education (HE) group received mailed materials (typically 1-2 pages) every 3 months. This included general information on Alzheimer's and dementia risk reduction using materials from sources such as the Alzheimer's Association and educational materials commonly provided as part of routine care at Kaiser Permanente Washington (KPWA).
Period: Overall Study
Arm/Group | SMARRT Intervention | Health Education Control
Started | 82 | 90
Completed | 68 | 81
Not Completed | 14 | 9
Not completed — Withdrawal by Subject | 4 | 8
Not completed — Lost to Follow-up | 7 | 0
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SMARRT Intervention | Health Education Control | Total
Number analyzed (Participants) | 82 | 90 | 172
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.8 (4.9) | 75.6 (4.6) | 75.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 51 | 108
  Male | 25 | 39 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 62 | 72 | 134
  Unknown or Not Reported | 18 | 13 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 8 | 17
  White | 64 | 68 | 132
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 4 | 4 | 8
Education, years [Mean (Standard Deviation); unit: years] — Years of formal education completed. For example, 12 years = High School Graduate.
  years | 16.0 (2.8) | 16.4 (2.4) | 16.2 (2.6)
Elixhauser comorbidity score [Mean (Standard Deviation); unit: units on a scale] — The Elixhauser Comorbidity Index (Elixhauser, 1998) is a risk score that measures the overall severity of comorbid illnesses (using diagnostic codes). Scores can range from 0 to 31. Higher scores represent higher severity of comorbid illnesses in the year prior to baseline and are associated with higher risk of mortality and hospital resource use.
  units on a scale | 2.8 (1.9) | 2.3 (1.7) | 2.5 (1.8)
Number of Risk Factors [Mean (Standard Deviation); unit: Risk Factors] — Average number of risk factors present at baseline, out of a total of 8 risk factors.
  Risk Factors | 2.5 (0.7) | 2.4 (0.6) | 2.5 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Change
Description: Cognitive function will be measured by the modified Neuropsychological Test Battery (mNTB) global score, which is a composite z-score, an average of z-scores from tests of several cognitive domains. The total score is reported. Higher values signify higher cognitive performance. A z-score of 0 represents the population mean.
  Treatment effects were estimated using linear mixed models (LMMs) for the changes from baseline to each follow-up assessment (6, 12, 18, and 24 months), with average treatment effects (ATEs) estimated by the average of the four visit-specific between-group differences in adjusted mean change from baseline.
  Changes made to the protocol due to Covid-19, i.e., switching to telephone data collection, will likely limit our ability to examine cognitive change effectively, as several of the most important cognitive tests cannot be administered via telephone.
Time Frame: 2 Years
Population: Participants were all members of Kaiser Permanente Washington (KPWA), an integrated healthcare delivery system in the Seattle area. Eligible participants were KPWA members aged 70-89, who had at least two of the following dementia risk factors targeted by the intervention: physical inactivity, uncontrolled hypertension, poor sleep, taking a prescription medication that may adversely affect cognition, high depressive symptoms, uncontrolled diabetes, social isolation, and current smoking.
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | SMARRT Intervention | Health Education Control
Number analyzed (Participants) | 82 | 90
z-score | 0.34 [0.25 to 0.42] | 0.19 [0.11 to 0.26]
Statistical Analysis 1: Comparison: SMARRT Intervention vs Health Education Control; Test type: Superiority; p = 0.008, Mixed Models Analysis — Adjusted for baseline value, sex, race/ethnicity education, comorbidity score and phone assessment; Treatment effects were estimated using linear mixed models (LMMs) for the changes from baseline to each follow-up assessment; Mean Difference (Net) = 0.15, 95% CI 2-sided [0.04 to 0.26]

2. Secondary Outcome: Change in Targeted Risk Factors
Description: A composite Z-score for risk factors based on the following: the Rapid Assessment of Physical Activity for Older Adult (RAPA), steps per day averaged over 7 days; blood pressure measures averaged for each six-month period for participants with hypertension; the Pittsburgh Sleep Quality Index (PSQI); use of potentially harmful prescription medications; the Center for Epidemiologic Studies - Depression Scale (CES-D); hemoglobin A1c (HbA1c) values averaged over a 12-month time period; the Patient-Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Social Activities, Short Form; and self-reported smoking. Higher score indicates greater risk factor burden. A z-score of 0 represents the population mean.
  Treatment effects were estimated using LMMs for the changes from baseline to each follow-up assessment (6, 12, 18, and 24 months), with ATEs estimated by the average of the four visit-specific between-group differences in adjusted mean change from baseline.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: z-score
Arm/Group | SMARRT Intervention | Health Education Control
Number analyzed (Participants) | 82 | 90
z-score | 0.06 [-0.01 to 0.13] | -0.05 [-0.12 to 0.02]
Statistical Analysis 1: Comparison: SMARRT Intervention vs Health Education Control; Test type: Superiority; p = 0.002, Mixed Models Analysis — Adjusted for baseline value, sex, race/ethnicity education, comorbidity score and phone assessment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.11, 95% CI 2-sided [0.02 to 0.21]

3. Secondary Outcome: Quality of Life Measure
Description: Measured with Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health. Higher score indicates better global health and quality of life; range = 0 to 20.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SMARRT Intervention | Health Education Control
Number analyzed (Participants) | 82 | 90
score on a scale | 12.69 [9.44 to 15.93] | 11.58 [8.36 to 14.79]
Statistical Analysis 1: Comparison: SMARRT Intervention vs Health Education Control; Test type: Superiority; p = 0.03, Mixed Models Analysis — Adjusted for baseline value, sex, race/ethnicity education, comorbidity score and phone assessment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 1.11, 95% CI 2-sided [0.08 to 2.14]

4. Secondary Outcome: Number of Participants With Mild Cognitive Impairment, Alzheimer's Disease, and Dementia
Description: Number of participants at follow up visits with Mild Cognitive Impairment, Alzheimer's Disease, and/or Dementia or with a low score on the Cognitive Abilities Screening Instrument (CASI) (<27 consistent with cognitive impairment). Lower score indicates poorer cognition; range is 0-33.
Time Frame: 2 Years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SMARRT Intervention | Health Education Control
Number analyzed (Participants) | 82 | 90
Participants | 5 | 8
Statistical Analysis 1: Comparison: SMARRT Intervention vs Health Education Control; Test type: Superiority; p = 0.52, Fisher Exact — Adjusted for age and sex; In an exploratory outcome, we examined incidence of a low CASI score or a diagnosis of MCI or dementia by treatment group; Odds Ratio (OR) = 0.68, 95% CI 2-sided [0.19 to 2.19]

ADVERSE EVENTS:
Time Frame: 24 months
Description: 1. Main Ascertainment: All participants are asked to report hospitalizations, new serious medical conditions, and new serious disabilities every three months, via AE form. This constitutes systematic assessment.
  2. Additional Reporting: Participants randomized to the intervention arm report incidental AEs during their coaching visits and phone calls. This constitutes non-systematic assessment. All possibly related, non-serious AEs are listed.
  None of the SAEs are study related.
Arm/Group | SMARRT Intervention | Health Education Control
All-Cause Mortality (participants affected / at risk) | 3/82 | 1/90
Serious Adverse Events (participants affected / at risk) | 24/82 | 23/90
Other Adverse Events (participants affected / at risk) | 14/82 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMARRT Intervention (N=82) | Health Education Control (N=90)
Hospitalizations (Blood and lymphatic system disorders) | 1 | 0
Hospitalizations (Cardiac disorders) | 5 | 4
Hospitalizations (Gastrointestinal disorders) | 5 | 4
Hospitalizations (General disorders) | 2 | 0
Hospitalizations (Hepatobiliary disorders) | 1 | 0
Hospitalizations (Musculoskeletal and connective tissue disorders) | 3 | 2
Hospitalizations (Renal and urinary disorders) | 2 | 1
Hospitalizations (Reproductive system and breast disorders) | 1 | 0
Hospitalizations (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hospitalizations (Surgical and medical procedures) | 2 | 0
Life-Threatening Event (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hospitalizations (Endocrine disorders) | 0 | 1
Hospitalizations (Infections and infestations) | 0 | 3
Hospitalizations (Vascular disorders) | 0 | 5
Life-Threatening Event (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SMARRT Intervention (N=82) | Health Education Control (N=90)
Non-Serious, Possibly Related (Musculoskeletal and connective tissue disorders) | 9 | 0 — Calf cramps, joint pain, muscle pulls
Non-Serious, Possibly Related (Psychiatric disorders) | 2 | 0 — Study-related anxiety
Non-Serious, Possibly Related (Cardiac disorders) | 2 | 0 — High blood pressure at study visit
Non-serious, Possibly Related (Skin and subcutaneous tissue disorders) | 1 | 0 — Rash from activity monitor

LIMITATIONS AND CAVEATS:
Our trial was initiated prior to the COVID-19 pandemic, but the shutdown shortened the enrollment period and necessitated administering the intervention and measuring the outcomes remotely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/94/NCT03683394/Prot_SAP_000.pdf